CLINICAL TRIAL: NCT00991094
Title: Data Collection to Assess Acute and Late Normal Tissue Sequelae in Proton Therapy for Adults
Brief Title: Data Collection for the Assessment of Acute and Late Normal Tissue in Patients Treated With Proton Therapy
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PCR05-0207; NCI-2020-08092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PCR05-0207 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma; Esophageal Carcinoma; Genitourinary System Carcinoma; Head and Neck Carcinoma; Hematopoietic and Lymphoid Cell Neoplasm; Lung Carcinoma; Malignant Central Nervous System Neoplasm; Malignant Digestive System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Esophageal Neoplasms; Hematologic Neoplasms; Lung Neoplasms; Central Nervous System Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients undergoing standard of care proton therapy are assessed for toxicities weekly during proton treatment, then from 1 to 3 times up to 90 days from the start of treatment and annually thereafter. Patients also complete questionnaires over 15-20 minutes at baseline, weekly during treatment, and every 2 weeks during follow up for up to 3 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study collects information on the side effects of proton therapy and detailed information on the proton therapy treatment plan itself. This may help researchers develop methods to predict the risk of side effects for future patients and learn the long-term benefit of proton therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively collect data on acute and late toxicities (including second malignant neoplasms) in patients treated with proton therapy.

II. To collect and store the corresponding radiation dose distribution and imaging data in order to correlate normal tissue response with dose distribution.

SECONDARY OBJECTIVES:

I. To derive and refine dose-response relationships for normal tissue toxicity after proton therapy.

II. To document and compare symptom burden weekly during treatment and twice a month for 3 months after therapy, using the M.D. Anderson Symptom Inventory (MDASI).

OUTLINE:

Patients undergoing standard of care proton therapy are assessed for toxicities weekly during proton treatment, then from 1 to 3 times up to 90 days from the start of treatment and annually thereafter. Patients also complete questionnaires over 15-20 minutes at baseline, weekly during treatment, and every 2 weeks during follow up for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for radiation treatment with protons at UTMDACC are eligible for this protocol
* Patients must sign a study-specific consent form prior to study entry

Exclusion Criteria:

* Patients who are unable or unwilling to attend the required periodic follow-ups either at M.D. Anderson or at a different site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for radiation treatment with protons at University of Texas M. D. Anderson Cancer Center (UTMDACC)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-05-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities data in patients treated with proton therapy | Up to 90 days after end of treatment
  Data will be collected from all organs receiving non-negligible proton dose during treatment. For each acute normal-tissue endpoint considered, analyses will be performed using the maximum toxicity score per patient within the 90-day follow-up. Upon analysis, the distribution of observed toxicity scores for each acute normal-tissue endpoint will be reported.
Late toxicities data in patients treated with proton therapy | Starting 90 days or more after the end of radiotherapy
  Data will be collected from all organs receiving non-negligible proton dose during treatment. For each late normal-tissue endpoint considered, analyses will be performed using censored time-to-event data corresponding to specified levels of injury (e.g. time to a specific grade >= 2 late toxicity). The log-rank test will be used to compare event times in subgroups of patients with different dosimetric characteristics of treatment (e.g. portion of lung receiving > 20 Gy: <= 40% vs > 40%). In addition, normal-tissue complication probability models will be fitted to data corresponding to incidence of a late endpoint within a specified time frame, with analysis limited to patients having the specified follow-up (e.g. incidence of grade >= 2 late rectal bleeding within 2 years among patients followed for 2 years post-treatment).
Dose-response relationships for normal tissue toxicity after proton therapy | Up to 3 months after therapy
  Relevant dose-volume response models from the literature, such as the Lyman model, the parallel model, or the critical-element model will be fitted to the data when possible, and model parameter estimates reported. Confidence intervals for model parameter estimates will be derived using the profile-likelihood method.

SECONDARY OUTCOMES:
Symptom burden | Up to 3 months after therapy
  Will be documented and compared using the M.D. Anderson Symptom Inventory (MDASI). The initial analysis for symptom data will be primarily descriptive in nature, and will include frequencies, proportions, means, medians, standard deviations, ranges, interquartile ranges, confidence intervals for the means, and box and whisker plots. Potential differences in symptom development between patients and between treatment variables will be explored using longitudinal analysis performed with mixed models.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Frank, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gjyshi O, Xu T, Elhammali A, Boyce-Fappiano D, Chun SG, Gandhi S, Lee P, Chen AB, Lin SH, Chang JY, Tsao A, Gay CM, Zhu XR, Zhang X, Heymach JV, Fossella FV, Lu C, Nguyen QN, Liao Z. Toxicity and Survival After Intensity-Modulated Proton Therapy Versus Passive Scattering Proton Therapy for NSCLC. J Thorac Oncol. 2021 Feb;16(2):269-277. doi: 10.1016/j.jtho.2020.10.013. Epub 2020 Oct 22. PMID 33198942
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org